CLINICAL TRIAL: NCT00216905
Title: Neurobiological Correlates of Disturbed Cognitive Function in Patients With Alcoholism - Simultaneous Measurement With EEG and fMRI
Brief Title: Simultaneous Measurement of Electroencephalography (EEG) and Functional Magnetic Resonance Imaging (fMRI) in Patients With Alcoholism
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: C. Mulert, MD, University of Munich
Other Study IDs: Mulert_LMU_EEG/fMRI; EK166/02
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Alcoholism
Keywords: Patients with alcoholism according to ICD-10 after detoxification
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Investigation of inpatients with alcoholism after detoxification with simultaneous Electroencephalography (EEG) and functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or more
* Inpatient with alcoholism after detoxification.

Exclusion Criteria:

* Neurological disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with alcohol use disorder
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mulert, M.D., Principal Investigator — Department of Psychiatry, Ludwig-Maximilians-University
Locations (1):
- Department of Psychiatry, Ludwig-Maximilians-University, Munich, Bavaria, Germany